CLINICAL TRIAL: NCT07310979
Title: Biomechanical and Clinical Effects of a Hyperbolic Paraboloid Triple-Abutment System on Morse Taper Dental Implants: Prospective Clinical Study With Finite Element Corroboration
Brief Title: Clinical Evaluation of a Hyperbolic Paraboloid Triple-Abutment on Morse Taper Dental Implants
Status: Enrolling by invitation | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Fernando O Costa, Titular professor, Federal University of Minas Gerais
Other Study IDs: 5957583
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Dental Implants; Dental Prosthesis, Implant-Supported
Keywords: Abutment design; Dental Implants; Biomechanics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Triple-Abutment System with Hyperbolic Paraboloid Geometry — Prosthetic loading will be performed on osseointegrated morse taper dental implants using a fixed implant-supported rehabilitation with a triple-abutment system featuring hyperbolic paraboloid geometry. Metal-ceramic prostheses will be cemented over the abutment components. All procedures will be performed by a single operator.

SUMMARY:
This prospective clinical study aims to evaluate the clinical and radiographic outcomes of a novel triple-abutment system with hyperbolic paraboloid geometry installed on Morse taper dental implants. The system is designed to support three adjacent crowns on a single implant, aiming to optimize load distribution and preserve peri-implant tissue stability.

Thirty systemically healthy adults missing three adjacent teeth will undergo implant placement, followed by a healing period of approximately three months for osseointegration prior to prosthetic loading. Metal-ceramic restorations will then be cemented over triple abutments. Clinical and radiographic evaluations will be performed at T1 (3-4 months after prosthetic loading) and T2 (12-18 months after prosthetic loading).

The primary outcome will be marginal bone level change assessed by standardized periapical radiographs. Secondary outcomes include probing depth, bleeding on probing, plaque index, keratinized mucosa height, and patient-reported satisfaction. The study aims to investigate whether this innovative abutment design provides stable peri-implant conditions and favorable clinical performance when applied to Morse taper implants.

DETAILED DESCRIPTION:
This prospective clinical study aims to evaluate the clinical and radiographic performance of an innovative triple-abutment (TA) system with hyperbolic paraboloid geometry installed on Morse taper dental implants. The abutment system is designed to support three adjacent crowns on a single implant through a fully curved, passive, non-welded configuration, with the objective of optimizing biomechanical load distribution and preserving peri-implant tissue stability. The concept is based on principles of mechanobiology, mechanotransduction, and biotensegrity, integrated within the framework of Optimized Biodynamic Peri-Implant Tissue (BOPiT).

Thirty systemically healthy adult participants presenting with three adjacent missing teeth will be enrolled. Implant placement will be performed following conventional surgical protocols. After surgery, a healing period of approximately three months will be allowed to achieve osseointegration prior to prosthetic loading. Subsequently, metal-ceramic fixed prostheses will be cemented over triple-abutment components. All surgical and prosthetic procedures will be conducted by a single experienced operator to ensure standardization.

Clinical and radiographic evaluations will be performed at two predefined follow-up timepoints: T1, corresponding to 3-4 months after prosthetic loading, and T2, corresponding to 12-18 months after prosthetic loading. The primary outcome measure will be marginal bone level change, assessed on standardized periapical radiographs obtained using the parallel technique with controlled calibration, and measured at the mesial and distal aspects of each implant.

Secondary outcome measures will include probing depth, bleeding on probing, plaque index, keratinized mucosa height, and patient-reported satisfaction assessed using a visual analog scale (VAS). Clinical maintenance visits will be scheduled every four months between T1 and T2 to monitor peri-implant health and prosthetic performance.

Statistical analyses will be conducted using parametric methods appropriate for repeated measures, with strategies to account for potential within-subject correlation in participants receiving more than one implant. Adverse events and biological or prosthetic complications will be recorded throughout the study period. The risks associated with participation are minimal and comparable to those of conventional implant-supported rehabilitations. In the event of complications, the triple-abutment system may be replaced by conventional abutments according to clinical judgment.

This study seeks to provide clinical evidence regarding the biomechanical and biological behavior of the triple-abutment system when applied to Morse taper implants, potentially supporting a more conservative and cost-effective rehabilitative approach by enabling the restoration of three adjacent teeth with a single implant while maintaining peri-implant tissue stability.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years.
* Systemically healthy as determined by medical history and clinical assessment.
* Non-smokers (no tobacco use).
* Able and willing to comply with study visits and maintenance program, and provide written informed consent.

Exclusion Criteria:

* diabetes mellitus (any type) or uncontrolled systemic disease.
* current or recent tobacco/nicotine use
* bisphosphonates or other antiresorptives,
* immunosuppressive therapy,
* osteoporosis
* pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample will be composed of adult patients with three adjacent missing teeth who underwent placement of a Morse taper dental implant, followed by a healing period of approximately three months for osseointegration. After confirmation of osseointegration, participants will be eligible for fixed implant-supported rehabilitation using a triple-abutment system designed to support a three-unit prosthesis on a single implant, according to clinical planning.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Changes in Marginal Bone Level (mm) | baseline vs. 3 months
  Marginal bone level measured in millimeters at the mesial and distal aspects of each implant using standardized periapical radiographs with the parallel technique and calibrated measurements, assessed at T1 (3-4 months)

SECONDARY OUTCOMES:
Changes in Marginal Bone Level (mm) | baseline vs. 12-18 months after prosthetic loading
  Marginal bone level measured in millimeters at the mesial and distal aspects of each implant using standardized periapical radiographs, assessed to evaluate medium-term peri-implant bone stability (12-18 months).
Changes in Peri-Implant Probing Depth | baseline versus 3-4 months (T2) after prosthetic loading
  Probing depth measured in millimeters at six sites per implant using a standardized periodontal probe.
Changes in Peri-Implant Probing Depth | baseline versus 12-18 months (T2) after prosthetic loading
  Probing depth measured in millimeters at six sites per implant using a standardized periodontal probe.
Presence of Bleeding on Probing | baseline versus 3-4 months (T2) after prosthetic loading
  Presence or absence of bleeding on probing assessed at six peri-implant sites per implant and expressed as the percentage of sites with bleeding.
Presence of Bleeding on Probing | baseline versus 12-18 months (T2) after prosthetic loading
  Presence or absence of bleeding on probing assessed at six peri-implant sites per implant and expressed as the percentage of sites with bleeding.
Presence of dental plaque | baseline versus 3-4 months (T2) after prosthetic loading
  Presence of dental plaque assessed at peri-implant sites and expressed as the percentage of sites with visible plaque.
Presence of dental plaque | baseline versus 12-18 months (T2) after prosthetic loading
  Presence of dental plaque assessed at peri-implant sites and expressed as the percentage of sites with visible plaque.
Changes in Keratinized Mucosa Height | baseline versus 3-4 months (T2) after prosthetic loading
  Width of keratinized peri-implant mucosa measured in millimeters at the mid-buccal aspect of each implant.
Changes in Keratinized Mucosa Height | baseline versus 12-18 months (T2) after prosthetic loading
  Width of keratinized peri-implant mucosa measured in millimeters at the mid-buccal aspect of each implant.
Level of Patient Satisfaction | baseline versus 3-4 months (T2) after prosthetic loading
  Patient-reported satisfaction with the implant-supported prosthetic rehabilitation assessed using a visual analog (VAS) scale. VAS ranging from 0 to 10; 10 indicates a complete satisfaction score.
Level of Patient Satisfaction | baseline versus 12-18 months (T2) after prosthetic loading
  Patient-reported satisfaction with the implant-supported prosthetic rehabilitation assessed using a visual analog (VAS) scale. VAS ranging from 0 to 10; 10 indicates a complete satisfaction score.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando O Costa, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Dental School, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.